CLINICAL TRIAL: NCT00003784
Title: A Phase II Pilot Trial of CHOP Followed by Iodine-131-Labeled Monoclonal Anti-B1 Antibody for Treatment of Newly Diagnosed Follicular Non-Hodgkin's Lymphomas
Brief Title: S9911, Combination Chemotherapy Plus Monoclonal Antibody Therapy in Treating Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066917; S9911 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-08-04 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Lymphoma
Keywords: Waldenström macroglobulinemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia; Lymphoma, Follicular | interventions — VAP-cyclo protocol; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine; tositumomab I-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CHOP regimen
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate
Radiation: tositumomab and iodine I 131 tositumomab

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by monoclonal antibody therapy in treating patients who have newly diagnosed follicular non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the 2 year failure free survival rate of patients with newly diagnosed follicular lymphoma treated with cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) followed by iodine I 131 monoclonal antibody anti-B1. II. Determine the complete and partial response rates of these patients after this therapy. III. Evaluate the toxicity of this regimen in these patients. IV. Determine the rate of disappearance of cells with clonal t(14;18)/bcl2 rearrangements from the peripheral blood and bone marrow after this therapy in these patients.

OUTLINE: Patients receive cyclophosphamide IV over 15 minutes, doxorubicin IV, and vincristine IV on day 1 and oral prednisone on days 1-5. Treatment is repeated every 21 days for up to 6 courses. Within 4-8 weeks after the last course of chemotherapy, patients who achieve at least a partial response and have less than 25% bone marrow involvement begin immunotherapy. Patients receive unlabeled monoclonal antibody anti-B1 (MOAB anti-B1) IV over 1 hour, then iodine I 131 MOAB anti-B1 IV over 20 minutes on day 1. This regimen is repeated on day 8. Patients are followed every 6 months for 2 years, then annually thereafter.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed follicular non-Hodgkin's lymphoma No prior treatment Bulky stage II, stage III, or stage IV Must express cluster of differentiation antigen 20 (CD20) antigen Bidimensionally measurable disease No Central Nervous System (CNS) involvement

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: Granulocyte count at least 1500/mm3 Platelet count at least 100,000/mm3 Hepatic: Not specified Renal: Not specified Cardiovascular: No arrhythmias (except sinus arrhythmia or infrequent premature ventricular contractions) No history of impaired cardiac status (severe coronary artery disease, cardiomyopathy, congestive heart failure, or serious arrhythmia Ejection fraction at least normal Other: HIV negative No prior malignancy within past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix No pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior monoclonal antibodies Chemotherapy: No prior chemotherapy for lymphoma Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy for lymphoma Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 1999-05; Primary Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver W. Press, MD, PhD, Study Chair — University of Washington
Locations (87):
- United States (87):
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Beckman Research Institute, City of Hope, Duarte, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Hospital - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Background] Hsi ED, Rimsza L, Goldman BH, et al.: MUM1 expression in follicular lymphoma is a poor prognostic marker in patients treated with immunochemotherapy (SWOG 9800/9911) but not chemotherapy alone (SWOG 8809): a Southwest Oncology Group correlative science study. [Abstract] Blood 112 (11): A-376, 2008.
- [Background] Fisher RI, LeBlanc M, Press OW, Maloney DG, Unger JM, Miller TP. New treatment options have changed the survival of patients with follicular lymphoma. J Clin Oncol. 2005 Nov 20;23(33):8447-52. doi: 10.1200/JCO.2005.03.1674. Epub 2005 Oct 17. PMID 16230674
- [Result] Press OW, Unger JM, Braziel RM, Maloney DG, Miller TP, Leblanc M, Fisher RI; Southwest Oncology Group. Phase II trial of CHOP chemotherapy followed by tositumomab/iodine I-131 tositumomab for previously untreated follicular non-Hodgkin's lymphoma: five-year follow-up of Southwest Oncology Group Protocol S9911. J Clin Oncol. 2006 Sep 1;24(25):4143-9. doi: 10.1200/JCO.2006.05.8198. Epub 2006 Aug 8. PMID 16896003
- [Result] Press OW, Unger J, Maloney D, et al.: An update of a phase II trial of CHOP followed by tositumomab/iodine I-131 tositumomab (Bexxar®) for front-line treatment of advanced stage, follicular lymphoma: Southwest Oncology Group Protocol 9911. [Abstract] Blood 106 (11): A-352, 2005.
- [Result] Press OW, Unger JM, Braziel RM, Maloney DG, Miller TP, LeBlanc M, Gaynor ER, Rivkin SE, Fisher RI. A phase 2 trial of CHOP chemotherapy followed by tositumomab/iodine I 131 tositumomab for previously untreated follicular non-Hodgkin lymphoma: Southwest Oncology Group Protocol S9911. Blood. 2003 Sep 1;102(5):1606-12. doi: 10.1182/blood-2003-01-0287. Epub 2003 May 8. PMID 12738671
- [Result] Press OW, Unger JM, Braziel RM, et al.: A phase II trial of CHOP followed by Bexxar™ (tositumomab and iodine-131-tositumomab) for treatment of newly diagnosed follicular non-Hodgkin's lymphomas (SWOG 9911). [Abstract] Blood 98 (11 Pt 1): A-3504, 2001.